CLINICAL TRIAL: NCT04816812
Title: The IBD-FITT Study - Moderate-intensity Exercise for Patients With Inflammatory Bowel Disease With Moderate Disease Activity: a Randomized Controlled Trial
Brief Title: The IBD-FITT Study - Moderate-intensity Exercise for IBD Patients With Moderate Disease Activity
Acronym: IBD-FITT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Ken Lund, Principal Investigator, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IBD-FITT_1
Record Dates: First submitted 2021-03-19; First posted 2021-03-25 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-12

CONDITIONS: Inflammatory Bowel Diseases
Keywords: Exercise
MeSH Terms: conditions — Inflammatory Bowel Diseases; Motor Activity

STUDY DESIGN:
Intervention Model Description: The investigators will apply a superior trial design in this randomized clinical trial with two arms, intervention, and comparison.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Other): In the intervention arm, a 12-week aerobic exercise program tailored to the individual patients by physiotherapists using the principles of Frequency, Intensity, Time, and, Type (FITT) aiming to increase or maintain the physical activity level to a weekly moderate activity level.
  Interventions: Behavioral: Exercise intervention; Behavioral: Lifestyle - online lesson intervention
- Comparison (Other): Comparison
  Interventions: Behavioral: Lifestyle - online lesson intervention

INTERVENTIONS:
Behavioral: Exercise intervention — A 12-week aerobic exercise program tailored to the individual patients by physiotherapists using the principles of Frequency, Intensity, Time, and, Type (FITT) aiming to increase or maintain the physical activity level to a weekly moderate activity level. This includes two supervised exercise sessions of 60 minutes per week, combined with one weekly home training session. The type of exercise is planned by a physiotherapist to fit each patient during sessions. We monitor the intervention by training diaries including frequency, intensity, time, and type of exercise (FITT) and the verbal BORG 15-point scale and heart rate monitors. We will also monitor the overall seven days' physical activity level by accelerometry using the AX3 device from the company Axivity at weeks 0 and 12.
  Arms: Exercise
Behavioral: Lifestyle - online lesson intervention — The investigators offer one online lesson of 15-25 minutes on lifestyle guidance including general advice on healthy living.

SUMMARY:
The investigators aim to investigate whether exercise therapy during 12 weeks including a lesson on general healthy lifestyle in adult patients with a moderately active disease is more effective, compared to control patients only receiving a lesson on general healthy lifestyle recommendations. The three main categories of outcomes are 1) health-related quality of life, 2) general health status of the patients 3) explorative outcomes. The primary outcome is health-related quality of life, the secondary outcome is general health status measured by waist circumference, disease activity scores, blood pressure, and blood lipids, and the third outcome are explorative outcomes (none-disease specific quality of life scores, biomarkers of C-reactive protein, fecal calprotectin and immunology markers including interleukins).

DETAILED DESCRIPTION:
The investigators will apply a superior trial design in this randomized clinical trial with two arms, intervention and comparison. In both the intervention and comparison arm, the patients will receive the proper and usual medical treatment decided by their responsible physician and changes in the medical treatment is allowed at all times.

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderately active Crohn's disease or ulcerative colitis are defined by fulfilling all the following five criteria:

  1. Well-characterized Crohn's disease or ulcerative colitis (physician assessment) i. Fulfilling standard clinical, endoscopic, radiologic, and histological criteria
  2. A minimum of one-year disease duration from the time of diagnosis of Crohn's disease or ulcerative colitis to inclusion into the trial
  3. Any of the following pharmacological treatments in a period of three months prior to inclusion:

     i. Usage of 5-Aminosalicylic acid (5-ASA) ii. Usage of corticosteroids iii. Immunomodulators usage: Azathioprine (AZA), 6-mercaptopurine (6-MP), Methotrexate (MTX) iv. Biologics usage: Anti-TNFα (Infliximab, Adalimumab, Golimumab), Ustekinumab or Anti-integrin (Vedolizumab)
  4. Disease activity defined by clinical disease score:

     i. Harvey Bradshaw Index (HBI) 27 > 5 ii. Simple Clinical Colitis Activity Index (SCCAI) 29 > 5
  5. Marker for gastrointestinal inflammation:

     i. Fecal calprotectin (FC) > 200 mg/g

     Exclusion Criteria:
* 1. A language barrier that prohibits the exercise instructors/supervisors to give sufficient or safe instructions during the intervention or at the general health lesson.

  2. Known heart condition that prevents them to actively participate safely in the exercise intervention.

  3. Known pregnancy or planned pregnancy. 4. Disabling musculoskeletal injuries that prevent them to actively participate in the exercise intervention.

  5. Severe disease activity manifested clinically and with the need for urgent change in treatment evaluated by the responsible physician.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Inflammatory Bowel Disease Questionnaire (IBDQ) | 12 weeks
  Health-related quality of life

SECONDARY OUTCOMES:
General health - Waist circumference | 12 weeks
  Waist circumference
General health - blood pressure | 12 weeks
  Blood pressure
General health - Lipid | 12 weeks
  Lipid status:
  i. Low-density lipoprotein (LDL) ii. High-density lipoprotein (HDL) iii. Triglycerides iv. Total cholesterol v. Hemoglobin A (Hbac1)
General health - Clinical disease activity | 12 weeks
  Harvey Bradshaw Index (Crohn's disease) Simple Clinical Colitis Activity Index (Ulcerative colitis)

OTHER OUTCOMES:
Explorative - European Quality of life | 12 weeks
  European Quality of life (EQ5D)
Explorative - Biomarkers | 12 weeks
  i. Fecal calprotectin ii. C-reactive protein iii. Immunology (cytokines)

CONTACTS AND LOCATIONS:
Overall Officials: Ken Lund, PhD, Principal Investigator — Odense University Hospital & University of Southern Denmark
Locations (2):
- Denmark (2):
  - Hospital of Southwest Jutland, Esbjerg
  - Odense University Hospital, Odense

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Elia J, Kane S. Adult Inflammatory Bowel Disease, Physical Rehabilitation, and Structured Exercise. Inflamm Bowel Dis. 2018 Nov 29;24(12):2543-2549. doi: 10.1093/ibd/izy199. PMID 29850914
- [Background] Shephard RJ. The Case for Increased Physical Activity in Chronic Inflammatory Bowel Disease: A Brief Review. Int J Sports Med. 2016 Jun;37(7):505-15. doi: 10.1055/s-0042-103157. Epub 2016 Apr 26. PMID 27116344
- [Background] Eckert KG, Abbasi-Neureither I, Koppel M, Huber G. Structured physical activity interventions as a complementary therapy for patients with inflammatory bowel disease - a scoping review and practical implications. BMC Gastroenterol. 2019 Jul 2;19(1):115. doi: 10.1186/s12876-019-1034-9. PMID 31266461
- [Background] Bilski J, Mazur-Bialy A, Brzozowski B, Magierowski M, Zahradnik-Bilska J, Wojcik D, Magierowska K, Kwiecien S, Mach T, Brzozowski T. Can exercise affect the course of inflammatory bowel disease? Experimental and clinical evidence. Pharmacol Rep. 2016 Aug;68(4):827-36. doi: 10.1016/j.pharep.2016.04.009. Epub 2016 May 2. PMID 27255494
- [Background] Reed JL, Pipe AL. Practical Approaches to Prescribing Physical Activity and Monitoring Exercise Intensity. Can J Cardiol. 2016 Apr;32(4):514-22. doi: 10.1016/j.cjca.2015.12.024. Epub 2015 Dec 29. PMID 26897182
- [Background] Bandholm T, Christensen R, Thorborg K, Treweek S, Henriksen M. Preparing for what the reporting checklists will not tell you: the PREPARE Trial guide for planning clinical research to avoid research waste. Br J Sports Med. 2017 Oct;51(20):1494-1501. doi: 10.1136/bjsports-2017-097527. Epub 2017 Sep 7. No abstract available. PMID 28882839
- [Derived] Lund K, Knudsen T, Kjeldsen J, Nielsen RG, Juhl CB, Norgard BM. The IBD-FITT study - moderate-intensity exercise for patients with inflammatory bowel disease with moderate disease activity: an open-label randomized controlled trial. Trials. 2023 Nov 20;24(1):742. doi: 10.1186/s13063-023-07781-4. PMID 37986021